CLINICAL TRIAL: NCT02867241
Title: An Intervention to Protect Young Children From Tobacco Smoke Exposure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laura J. Rosen (Other)
Collaborators: Flight Attendant Medical Research Institute (FAMRI) (Unknown); Hebrew University (Unknown); Assaf-Harofeh Medical Center (Other Government); Tel Aviv University (Other)
Responsible Party: Sponsor-Investigator, Laura J. Rosen, Senior Lecturer and Chair, Dept. of Health Promotion, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0143-16ASF
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Passive Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): 1. Motivational interviews (3 visits) + supportive phone calls
  2. Feedback of child hair nicotine levels
  3. Feedback of home air quality (PM2.5)
  4. New Media (Website and/or Facebook with information and parental forum)
  Interventions: Behavioral: Behavioral Early
- Control Regular (Other): This group will get no intervention during the study period. Following the close of the study, participants in this group will receive a shortened version of the intervention (1 motivational interview, with feedback on child hair nicotine levels and feedback on home air quality (PM2.5))
  Interventions: Behavioral: Behavioral Late
- Control Expanded (Other): This group will get no intervention during the study period. However, participants will fill out a detailed questionnaire on parental perceptions of exposure and risk, as well as questions on social norms, self-efficacy, and knowledge Following the close of the study, participants in this group will receive a shortened version of the intervention (1 motivational interview, with feedback on child hair nicotine levels and feedback on home air quality (PM2.5))
  Interventions: Behavioral: Behavioral Late

INTERVENTIONS:
Behavioral: Behavioral Early — Participants will receive an intervention which includes motivational interviewing, biochemical feedback, air quality feedback, phone calls, and social media
  Arms: Intervention
Behavioral: Behavioral Late — After the close of the study, Participants will receive an intervention which includes motivational interviewing, biochemical feedback, air quality feedback, phone calls, and social media
  Arms: Control Expanded; Control Regular

SUMMARY:
The primary goal of this research is to evaluate the effectiveness of an intervention for parents to reduce tobacco smoke exposure of young children

DETAILED DESCRIPTION:
The primary aim of this intervention is to reduce exposure of children to tobacco smoke, through an intervention program designed to help parents better perceive exposure and its harms, and to provide tools for assisting them in protecting children. Secondary aims are to understand the relationships between parentally-reported and objectively measured child tobacco smoke exposure, to assess the relationship between tobacco smoke exposure and health and health care utilization, and to better understand parental perceptions of tobacco smoke exposure (PPE) and parental perceptions of risk (PPR) from tobacco smoke exposure. The effectiveness of the intervention will be evaluated using a randomized controlled trial.

This RCT is a continuation of previous work. Originally the entire research project, which included a Pilot Study and a Randomized Controlled Trial (RCT) was registered as NCT01335178. Upon completion of the Pilot Study, we closed NCT01335178 and opened a new one for the RCT with the current registration number.

ELIGIBILITY:
Inclusion Criteria for RCT :

1. - Families in which at least one parent smokes, and both parents combined smoke a minimum of 10 cigarettes per week
2. - Parents willing to provide child hair samples
3. - Hebrew speaking participants
4. - Parents are willing to participate from time of entry for the coming 8 months .

Exclusion Criteria:

There are no additional exclusion criteria

-

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in child exposure to tobacco smoke as assessed by log hair nicotine | Baseline and 6 months post-enrollment
  A small amount of hair will be taken from the child's head near the scalp and sent to a laboratory for analysis

SECONDARY OUTCOMES:
Change in child exposure to tobacco smoke as assessed by parental report | Baseline and 6 months post-enrollment
  Frequency of child exposure to tobacco smoke as measured by a single question
Change in smoking practices in the home as reported by parents | Baseline and 6 months post-enrollment
  Smoking practices in the home as measured by a single question
Change in parental smoking | Baseline and 6 months post-enrollment
  Parental quit rates
Change in parental perceptions of risk due to smoking, intervention and expanded control groups | Baseline and 6 months post-enrollment
  Measurement of risk resulting in a single composite number using a validated questionnaire
Change in parental perceptions of tobacco smoke exposure, intervention and expanded control groups | Baseline and 6 months post-enrollment
  Measurement of exposure perceptions resulting in a single composite number using a validated questionnaire
Child health | 6 months post-enrollment
  Number of child illnesses related to tobacco smoke exposure
Child health services utilization | 6 months post-enrollment
  Number of visits to physicians or emergency care services
Change in smoking practices in the car as reported by parents | Baseline and 6 months post-enrollment
  Frequency of smoking in the car (single question)
Change in parentally-reported number of cigarettes smoked | Baseline and 6 months post-enrollment
  Reported number of cigarettes smoked by parents daily
Change in parentally-reported child exposure to tobacco smoke, intervention and expanded control groups | Baseline and 6 months post-enrollment
  Detailed parental report on when and how often child is exposed to tobacco smoke, as summarized by composite scale
Parental perceptions of risk due to smoking, intervention versus control group | 6 months post-enrollment
  Measurement of risk perceptions resulting in a single composite number using a validated questionnaire
Parental perceptions of tobacco smoke exposure, intervention versus control group | 6 months post-enrollement
  Measurement of exposure perceptions resulting in a single composite number using a validated questionnaire
Correlations between parentally-reported exposure and child log hair nicotine | baseline
  Pearson correlations
Correlations between parentally-reported exposure and child log hair nicotine | 6 months
  Pearson correlations

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Rosen, PhD, Principal Investigator — Tel Aviv University; David M Zucker, PhD, Study Director — Hebrew University
Locations (1):
- Tel Aviv University, Ramat Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosen L, Zucker D, Guttman N, Brown N, Bitan M, Rule A, Berkovitch M, Myers V. Protecting Children From Tobacco Smoke Exposure: A Randomized Controlled Trial of Project Zero Exposure. Nicotine Tob Res. 2021 Nov 5;23(12):2003-2012. doi: 10.1093/ntr/ntab106. PMID 34021353
- [Derived] Myers V, Shiloh S, Zucker DM, Rosen LJ. Changing Exposure Perceptions: A Randomized Controlled Trial of an Intervention with Smoking Parents. Int J Environ Res Public Health. 2020 May 12;17(10):3349. doi: 10.3390/ijerph17103349. PMID 32408551